CLINICAL TRIAL: NCT00453310
Title: A Phase II Study of Sunitinib in Patients With Refractory or Relapsed Germ Cell Tumors
Brief Title: Sunitinib in Treating Patients With Metastatic Germ Cell Tumors That Have Relapsed or Not Responded to Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-004; P30CA008748 (NIH); MSKCC-07004
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Results first posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-09

CONDITIONS: Extragonadal Germ Cell Tumor; Ovarian Cancer; Teratoma; Testicular Germ Cell Tumor
Keywords: recurrent ovarian germ cell tumor; stage IV ovarian germ cell tumor; ovarian choriocarcinoma; ovarian immature teratoma; ovarian mature teratoma; recurrent malignant testicular germ cell tumor; testicular choriocarcinoma; testicular seminoma; testicular yolk sac tumor; ovarian dysgerminoma; ovarian embryonal carcinoma; ovarian yolk sac tumor; ovarian monodermal and highly specialized teratoma; ovarian polyembryoma; stage III malignant testicular germ cell tumor; ovarian mixed germ cell tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and seminoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and yolk sac tumor; testicular embryonal carcinoma and seminoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular yolk sac tumor and teratoma with seminoma; testicular yolk sac tumor and teratoma; testicular embryonal carcinoma; recurrent extragonadal non-seminomatous germ cell tumor; recurrent extragonadal seminoma; stage IV extragonadal non-seminomatous germ cell tumor; stage IV extragonadal seminoma; recurrent extragonadal germ cell tumor; testicular immature teratoma; testicular mature teratoma; adult teratoma
MeSH Terms: conditions — Ovarian Neoplasms; Teratoma; Testicular Germ Cell Tumor; Testicular Neoplasms; Seminoma; Endodermal Sinus Tumor; Dysgerminoma; Carcinoma, Embryonal | interventions — Sunitinib

ARMS (1):
- sunitinib malate (Experimental): The dose of sunitinib malate will be a continuous daily dose of 37.5 mg administered orally for 6 weeks. The cycle of therapy is 42 days (or 6 weeks)
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sunitinib works in treating patients with metastatic germ cell tumors that have relapsed or not responded to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of sunitinib malate in patients with refractory or relapsed metastatic germ cell tumors.

Secondary

* Determine the safety of this drug in these patients.
* Determine the time to tumor response and duration of tumor response in patients treated with this drug.

OUTLINE: This is a open-label study.

Patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 6 weeks for up to 9 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed at 28 days and then periodically thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed seminoma or nonseminoma germ cell tumors (GCT)

  * Refractory or relapsed disease
  * Metastatic disease
* Progressive disease after prior cisplatin-based chemotherapy AND meets 1 of the following criteria for salvage therapy:

  * Not a candidate for potentially curative therapy
  * Received prior high-dose chemotherapy regimens
  * Declines potentially curative therapy (mediastinal GCT or primary refractory GCT)
* Measurable disease*, defined as 1 of the following:

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
  * Elevation of alpha-fetoprotein > 15 ng/mL and/or elevation of human chorionic gonadotropin > 2.2 mIU/L
* NOTE: *Patients with radiographically measurable disease only must have ≥ 1 site that has not undergone prior irradiation

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN (unless elevated liver function abnormalities due to underlying malignancy)
* LVEF ≥ 50% by MUGA
* No grade 3 hemorrhage within the past 4 weeks
* None of the following within the past 6 months:

  * Myocardial infarction
  * Severe or unstable angina
  * Coronary or peripheral artery bypass graft
  * Symptomatic congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Pulmonary embolism
* No prolonged QTc interval (i.e., QTc > 450 msec for males and > 470 msec for females)
* No ongoing cardiac dysrhythmias ≥ grade 2
* No uncontrolled hypertension, defined as blood pressure > 150/100 mm Hg despite optimal therapy
* No active infection
* No other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would preclude study compliance, according to the study investigator
* Not pregnant or nursing

  * Negative sonogram required to exclude pregnancy
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior sunitinib malate
* More than 4 weeks since prior major surgery and recovered
* More than 4 weeks since prior radiotherapy and recovered
* Concurrent palliative radiotherapy to metastatic lesion(s) allowed provided ≥ 1 measurable lesion has not been irradiated
* No concurrent therapeutic doses of warfarin

  * Low-dose oral warfarin (up to 2 mg daily) for prophylaxis and treatment or heparin products at prophylactic or treatment doses allowed
* No other concurrent investigational or approved anticancer therapies, including chemotherapy, biologic response modifiers, hormone therapy, or immunologic-based treatment

  * Concurrent participation in supportive care or nontreatment trials (e.g., quality-of-life or laboratory analyses) allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean F. Bajorin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Robert J. Motzer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Feldman DR, Turkula S, Ginsberg MS, Ishill N, Patil S, Carousso M, Bosl GJ, Motzer RJ. Phase II trial of sunitinib in patients with relapsed or refractory germ cell tumors. Invest New Drugs. 2010 Aug;28(4):523-8. doi: 10.1007/s10637-009-9280-2. Epub 2009 Jun 23. PMID 19547919

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib Malate: The dose of sunitinib malate will be a continuous daily dose of 37.5 mg administered orally for 6 weeks. The cycle of therapy is 42 days (or 6 weeks)
  sunitinib malate
Period: Overall Study
Arm/Group | Sunitinib Malate
Started | 10
Completed | 0
Not Completed | 10
Not completed — Progression of Disease | 10

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (Complete and Partial Response) as Measured by RECIST Criteria After 2 Courses of Treatment
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 10
participants
  Stable Disease | 3
  Progression of Disease | 7

ADVERSE EVENTS:
Arm/Group | Sunitinib Malate
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate (N=10)
Hemorrhage, Abdomen NOS (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate (N=10)
ALT, SGPT (Blood and lymphatic system disorders) | 2 (2)
Glucose, high (hyperglycemia) (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, Nose (General disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Mucositis (func/sympt)- Oral cavity (General disorders) | 2 (2)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Pain - Extremity-limb (General disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes